CLINICAL TRIAL: NCT05726409
Title: Mobile Application to Create Healthy Food Preparation Habits for Patients With Diabetes and Prediabetes: A Pilot Study
Brief Title: Mobile Application to Create Healthy Food Preparation Habits for Patients With Diabetes and Prediabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was never started due to lack of access to our proposed patient database.
Sponsor: Boston Medical Center (Other)
Collaborators: Boston Medical Center Food Kitchen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-42380
Record Dates: First submitted 2023-02-05; First posted 2023-02-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 2; Pre Diabetes
Keywords: Mobile application; Meal preparations; Recipes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile application user (Experimental): Each participant will be sent an email with a link to download a mobile application to access the meal planner function.
  Interventions: Other: Mobile application

INTERVENTIONS:
Other: Mobile application — Participants will use the meal planner function on the mobile application to plan and cook at least 3 meals a week for 12 weeks.

SUMMARY:
Boston Medical Center (BMC) serves many underserved, low-income patients and has developed an innovative strategy to combat food insecurity including a preventative food pantry, a teaching kitchen, and a rooftop farm that provides fresh produce directly to the patients. The presence of this well-established, three-pronged approach places BMC in an ideal position to develop a nutritional education intervention that supports experiential learning in this high-risk population.

For this first exploratory study, 75 enrolled participants will be given a free mobile application with recipes designed to build habits. Participants will cook at least three meals weekly for two months using the app. Self-reported survey data and activity on the app will be collected and used to assess the feasibility of teaching cooking skills through a mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Access to an oven OR microwave, stovetop OR hot plate, and food storage.
* Access to the internet on a smartphone
* Owns a smartphone with iOS Apple Store or Google Play
* Reading proficiency in English
* Has a diagnosis of diabetes or prediabetes(Hb A1C> 5.6)

Exclusion Criteria:

* Inability to provide informed consent
* Taking any medications or has a condition that limits the ability to increase intake of fruits and vegetables (including warfarin and end-stage renal disease)
* Attended a Diabetes Self-Management Education (DSME) at BMC within the past year or plans to attend during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of mobile app use | 12 weeks
  Data will be collected by the mobile app on the frequency of use throughout the 12 week intervention.
Recipe completion rate | 12 weeks
  Data will be collected by the mobile app on the rate of recipe completion throughout the 12 week intervention. Higher rates of completion are considered more favorable.
Satisfaction with the mobile application | 12 weeks
  An investigator developed satisfaction questionnaire will be used to assess satisfaction with the mobile application.

SECONDARY OUTCOMES:
Change in dietary patterns | baseline, 12 weeks
  This outcome will be measured using PrimeScreen, which is a validated brief dietary screening tool developed by the Harvard School of Public Health. It will provide the change in frequency of consumption of fruits, vegetables, lean protein, carbohydrates, fat, and processed foods.
Change in nutrition knowledge | baseline, 12 weeks
  Change in nutrition knowledge will be assessed through the adapted Slater Nutrition Knowledge Survey. These questions apply knowledge by asking participants to use their knowledge to make decisions rather than repeating the taught nutrition recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Ciszak, MD, Principal Investigator — Boston Medical Center, Department of Family Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No